CLINICAL TRIAL: NCT01440920
Title: A Phase I Study of OCV-501 in the Treatment of Patients With Acute Myeloid Leukemia
Brief Title: A Phase I Study of OCV-501 in Acute Myeloid Leukemia Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 311-10-001; JapicCTI-111623 (Other: JAPIC)
Record Dates: First submitted 2011-09-15; First posted 2011-09-27 (Estimated); Results first posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute myeloid leukemia; WT1
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): 0.3 mg
  Interventions: Drug: OCV-501
- Cohort 2 (Experimental): 1 mg
  Interventions: Drug: OCV-501
- Cohort 3 (Experimental): 3 mg
  Interventions: Drug: OCV-501

INTERVENTIONS:
Drug: OCV-501 — subcutaneously administered once a week, 4 times at the dose of 0.3 mg
  Arms: Cohort 1
Drug: OCV-501 — subcutaneously administered once a week, 4 times at the dose of 1 mg
  Arms: Cohort 2
Drug: OCV-501 — subcutaneously administered once a week, 4 times at the dose of 3 mg
  Arms: Cohort 3

SUMMARY:
The purpose of this study is to assess the safety, tolerability of OCV-501 in patients with acute myeloid leukemia (AML) who achieved complete remission after induction regimen and who completed a standard consolidation therapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients with acute myeloid leukemia including patients with secondary leukemia. However, the patients with MDS apparently evolved itno AML and patients with AML accompanied by t(15;17)(q22;q12),(PML/RARalpha) , should be excluded.
* Patients who achieved the first complete remission after the induction regimen and finished a standard consolidation therapy.
* Age: ≥ 60years of age(at the time of signature of the informed consent form)
* Sex: Male and Female
* Patients who are capable of giving informed consent
* Patient's blasts cells show expression of WT1mRNA, detected by quantitative RT-PCR.
* Patients must be one of the following HLA DRB1 types: HLA-DRB1*01:01, *04:05, *15:01, *15:02, *08:03 and *09:01.

Key Exclusion Criteria:

* Patients who are scheduled for a bone marrow transplantation
* Patients who were administered exceeded acceptable therapeutic dose of immunosuppressants and adrenal cortical steroids.
* Patients with uncontrollable active infectious diseases
* Patients with autoimmune diseases (including Hashimoto's disease, idiopathic thrombocytopenic purpura, and autoimmune hepatitis) or with a medical history of active autoimmune diseases
* Immunocompetent patients
* Patients with a complication of interstitial pneumonia or with a medical history of interstitial pneumonia

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-09; Primary Completion 2013-03 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center, Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: subcutaneously administered once a week, 4 times at the dose of 0.3 mg
- Cohort 2: subcutaneously administered once a week, 4 times at the dose of 1 mg
- Cohort 3: subcutaneously administered once a week, 4 times at the dose of 3 mg
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 3 | 3 | 3
Completed | 3 | 3 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1 | 2
  >=65 years | 2 | 3 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 0 | 4
  Male | 1 | 1 | 3 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 3 | 3 | 3 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 3 | 3 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Dose Limiting Toxicities
Description: Dose limiting toxicity (DLT) was defined as any of the following adverse events occurring by Day 29 (7 days after the last investigational medicinal product [IMP] administration) of this trial for which a causal relationship to the IMP could not be ruled out. Severity of the adverse events was evaluated in accordance with the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) ver. 4.0. Blood toxicity did not include hematology parameters of laboratory tests.
  * Non-blood toxicities ≥ Grade 3, excluding cases of anorexia, nausea, vomiting, diarrhea, and constipation where it is possible to continue the clinical trial by use of supportive therapy
  * Blood toxicities ≥ Grade 4, although febrile neutropenia ≥ Grade 3 will be counted as DLT.
Time Frame: 4 Weeks
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 3 | 3 | 3
participants | 0 | 0 | 0

2. Secondary Outcome: Recurrence Based on the Response Evaluation Criteria by the International Working Group
Description: A case will be designated as relapse if any of the following occur. Reappearance of leukemic blast cells in the peripheral blood or ≥5% blast cells in the bone marrow after complete remission (morphologic relapse).
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 3 | 3 | 3
participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from start of the first IMP administration (Day 1) to Post-treatment observation (Day 50).
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3) | Cohort 3 (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 1 | 0 | 0
Vitreous floaters (Eye disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Injection site erythema (General disorders) | 3 | 3 | 3
Injection site induration (General disorders) | 2 | 2 | 3
Injection site mass (General disorders) | 1 | 0 | 0
Injection site pain (General disorders) | 0 | 1 | 0
Injection site pruritus (General disorders) | 1 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Eosinophil count increased (Investigations) | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 1
Platelet count decreased (Investigations) | 1 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 1
Protein urine present (Investigations) | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No